CLINICAL TRIAL: NCT04061681
Title: Efficacy of Project BIPAMS for Restless Legs Syndrome in Adults With Multiple Sclerosis: A Pilot Study
Brief Title: Efficacy of BIPAMS for Restless Legs Syndrome in Adults With Multiple Sclerosis: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Robert W Motl, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003877
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis; Restless Legs Syndrome
Keywords: Physical Activity
MeSH Terms: conditions — Multiple Sclerosis; Restless Legs Syndrome; Motor Activity | interventions — Behavior Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions that will be occurring simultaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (BIPAMS) (Experimental): Participants will complete a 16-week behavioral intervention to increase physical activity levels.
  Interventions: Behavioral: Behavioral Intervention (BIPAMS)
- Waitlist Control (No Intervention): Participants will have 16-weeks of no intervention or interaction.

INTERVENTIONS:
Behavioral: Behavioral Intervention (BIPAMS) — This 16-week behavioral intervention teaches people the skills, techniques, and strategies based on Social Cognitive Theory of behavior change for modifying and self-regulating health behaviors, including physical activity. The behavioral intervention consists of two primary components, namely a dedicated Internet website and one-on-one video chats with a behavioral coach via SkypeTM.
  Other Names: Project BIPAMS: Behavioral Intervention for Physical Activity in Multiple Sclerosis (BIPAMS)
  Arms: Behavioral Intervention (BIPAMS)

SUMMARY:
The purpose of this study is to evaluate the efficacy of a 16-week behavioral intervention for increasing physical activity and reducing restless legs syndrome (RLS) severity in persons with multiple sclerosis (MS) and RLS. The study includes a proposed sample of 20 persons with MS and RLS that will be randomized into either a 16-week behavioral intervention arm aimed at increasing physical activity or a 16-week wait-list control arm.

DETAILED DESCRIPTION:
The primary aim of the proposed pilot RCT involves examining the efficacy of a 16-week behavioral intervention for increasing physical activity and reducing RLS severity in persons with MS and RLS. Secondarily, the investigators will be assessing changes in sleep quality and daytime sleepiness following the behavioral intervention. The study includes a proposed sample of 20 persons with MS and RLS that will complete a baseline testing session for measures of physical activity, restless legs syndrome severity, sleep quality, and daytime sleepiness. Participants will then be randomized into one of two study arms: (1) a 16-week Social Cognitive Theory-based behavioral intervention aimed at increasing physical activity; or (2) 16-week waitlist control with the option of completing the intervention upon completion of the study. All participants will complete a follow-up testing session at the conclusion of each 16-week arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* Relapse free in the past 30 days
* Positive screen for restless legs syndrome
* Non-active (not engaging in 30 minutes of activity per day on more than 2 days per week in the previous six months)
* Ambulatory without assistance
* Internet and email access

Exclusion Criteria:

* Diagnosis of radiculopathy, peripheral edema, peripheral neuropathy, iron deficiency (i.e., anemia) renal disease, or diabetes
* Screen at moderate or high risk for undertaking strenuous or maximal exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Restless Legs Syndrome Severity as measured by the International Restless Legs Syndrome Study Group Scale | Baseline
  Participants will complete the International Restless Legs Syndrome Study Group Scale (IRLS), a 10-item questionnaire that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life over the previous week.Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with total scores ranging from 0-40 and higher scores indicating a greater severity of symptoms.This will be completed at the baseline testing session.
Restless Legs Syndrome Severity as measured by the International Restless Legs Syndrome Study Group Scale | Follow-Up
  Participants will complete the International Restless Legs Syndrome Study Group Scale (IRLS), a 10-item questionnaire that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life over the previous week.Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with total scores ranging from 0-40 and higher scores indicating a greater severity of symptoms. This will be completed at the follow-up testing session.
Physical Activity Levels as measured by the Godin Leisure-Time Exercise Questionnaire | Baseline
  Participants will complete the Godin Leisure-Time Exercise Questionnaire (GLTEQ) as a measure of the frequency of strenuous, moderate, and mild leisure-time physical activity performed for periods of 15 minutes or more over a typical week. Summary scores are calculated by multiplying the number of strenuous, moderate, and mild bouts by 9, 5, and 3, respectively, and summing those values into an overall score that ranges from 0 to 119; higher scores are represent a greater volume of physical activity. This will be completed at baseline testing.
Physical Activity Levels as measured by the Godin Leisure-Time Exercise Questionnaire | Follow-Up
  Participants will complete the Godin Leisure-Time Exercise Questionnaire (GLTEQ) as a measure of the frequency of strenuous, moderate, and mild leisure-time physical activity performed for periods of 15 minutes or more over a typical week. Summary scores are calculated by multiplying the number of strenuous, moderate, and mild bouts by 9, 5, and 3, respectively, and summing those values into an overall score that ranges from 0 to 119; higher scores are represent a greater volume of physical activity. This will be completed at follow-up testing.

SECONDARY OUTCOMES:
Sleep Quality as measured by the Pittsburgh Sleep Quality Index | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) measures sleep quality and sleep disturbances over the past four weeks and containing seven different components of sleep. Components of sleep are scored from 0 (fairly good) to 3 (very bad) and component scores are summed for a global score ranging from 0-21; higher scores are indicative of worse sleep quality. Participants will complete this questionnaire at baseline testing.
Sleep Quality as measured by the Pittsburgh Sleep Quality Index | Follow-up
  The Pittsburgh Sleep Quality Index (PSQI) measures sleep quality and sleep disturbances over the past four weeks and containing seven different components of sleep. Components of sleep are scored from 0 (fairly good) to 3 (very bad) and component scores are summed for a global score ranging from 0-21; higher scores are indicative of worse sleep quality. Participants will complete this questionnaire at Follow-up testing.
Sleep Quality as measured by accelerometry | Baseline
  Accelerometry provides device-measured aspects of sleep quality including sleep onset latency, time in bed, total sleep time, frequency of awakenings, time awake after sleep onset, and sleep efficiency. Participants will be instructed to wear one ActiGraph GT3X+ accelerometer device on the non-dominant wrist each night (i.e., during time in bed for scheduled sleep time) for seven nights following the baseline testing session.
Sleep Quality as measured by accelerometry | Follow-up
  Accelerometry provides device-measured aspects of sleep quality including sleep onset latency, time in bed, total sleep time, frequency of awakenings, time awake after sleep onset, and sleep efficiency. Participants will be instructed to wear one ActiGraph GT3X+ accelerometer device on the non-dominant wrist each night (i.e., during time in bed for scheduled sleep time) for seven nights following the follow-up testing session.
Daytime Sleepiness as measured by the Epworth Sleepiness Scale | Baseline
  The Epworth Sleepiness Scale (ESS) is an 8-item questionnaire whereby participants are asked to rate how likely they would be to doze off or fall asleep during eight different situations in "recent times" to provide a global score of daytime sleepiness. Items are scored on a range of 0 (would never doze) to 3 (high chance of dozing) and summed to provide a global score of daytime sleepiness ranging between 0 and 24 with higher scores indicating more daytime sleepiness. Participants will complete the questionnaire at baseline testing.
Daytime Sleepiness as measured by the Epworth Sleepiness Scale | Follow-up
  The Epworth Sleepiness Scale (ESS) is an 8-item questionnaire whereby participants are asked to rate how likely they would be to doze off or fall asleep during eight different situations in "recent times" to provide a global score of daytime sleepiness. Items are scored on a range of 0 (would never doze) to 3 (high chance of dozing) and summed to provide a global score of daytime sleepiness ranging between 0 and 24 with higher scores indicating more daytime sleepiness. Participants will complete the questionnaire at Follow-up testing.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Motl, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cederberg KLJ, Motl RW. Feasibility and efficacy of a physical activity intervention for managing restless legs syndrome in multiple sclerosis: Results of a pilot randomized controlled trial. Mult Scler Relat Disord. 2021 May;50:102836. doi: 10.1016/j.msard.2021.102836. Epub 2021 Feb 10. PMID 33618120